CLINICAL TRIAL: NCT00239200
Title: Lapatinib (GW572016) a Dual Inhibitor of EGFR and ErbB2, for Metastatic or Recurrent Squamous Cell Carcinoma of the Esophagus
Brief Title: Lapatinib (GW572016) for Metastatic or Recurrent Squamous Cell Carcinoma Esophagus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: notification from sponsor
Sponsor: University of Michigan Rogel Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005-037
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Metastatic or Recurrent Squamous Cell Carcinoma of the Esophagus
MeSH Terms: conditions — Neoplasm Metastasis; Esophageal Squamous Cell Carcinoma | interventions — Lapatinib

INTERVENTIONS:
Drug: Lapatinib

SUMMARY:
The purpose of this study is the determine whether a new compound, called lapatinib, can be effective in shrinking cancerous tumors of the esophagus that have recurred or spread somewhere else in the body. They also want to determine the toxicity of this regimen. Lapatinib blocks 2 receptors that sometimes are present on cancer cells (called epidermal growth factor receptor, and the Erb B2 receptor). It is possible that blocking these receptors may decrease the growth of the cancer cells.

DETAILED DESCRIPTION:
The subject will take an oral pill called Lapatinib. Each tablet is 250 mg. Subjects will take 1500mg (six 250mg tablets) of lapatinib once daily. Subjects must fast 1 hour prior to and 1 hour following dosing. If a subject is unable to swallow lapatinib tablets whole, the lapatinib may be crushed with a mortar and pestle to form a powder, and mix it in 4 oz (120 ml) of water to take by mouth or through a feeding tube. Then the subject will then rinse the mortar with 2 oz (60ml) of water to suspend the left-over powder, and then swallow the rinse or flush it down the feeding tube. You will have to repeat this rinse one more time.

Subjects will have a "MUGA" scan done at the very beginning to make sure that heart function is good. It will then be repeated every other month while on treatment. When the subjects have a MUGA scan, 3 cc's (less than one teaspoon) of blood will be drawn from your vein, and labeled with a radioactive substance. Then, subjects blood will be injected back into his/her arm through a catheter in your vein. The level of radiation you will be exposed to is very minimal. Then, a camera will take a "movie" of your heart. The entire procedure lasts about 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic or recurrent squamous cell carcinoma of the esophagus.
* Patients must have histologically or cytologically confirmed disease.
* Patients may have received one prior regimen of neoadjuvant chemotherapy or chemoradiation, and prior esophagectomy is acceptable. Patients may also have received one prior chemotherapy regimen for recurrent disease.
* Patients may have received no more than 4500 cGy to fields including substantial marrow.
* Age greater than or equal than 18 years. Because no dosing or adverse event data are currently available on the use of GW572016 in patients <18 years of age, children are excluded from this study.
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

Leukocytes greater than or equal to 3,000/microliters Absolute neutrophil count greater than or equal to 1,500/microliters Platelets greater than or equal to 100,000/microliters Total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT)less than or equal to 2.5 X institutional upper limit of normal Creatine within normal institutional limits OR creatinine clearance greater than or equal to 60 ml/min for patients with creatinine levels above institutional normal

-Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan. A normal ejection fraction is equal or greater than 50%. Baseline and on treatment scans should be performed using the same modality and preferably at the same institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome:
Primary Objective: To determine the response rate of metastatic or recurrent squamous cell carcinoma of the esophagus, when treated with lapatinib (GW572016)

SECONDARY OUTCOMES:
Secondary Outcome:
Secondary Objective: To determine the toxicity of this regimen

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States